CLINICAL TRIAL: NCT01338714
Title: The Effect of Compound Herbal Formula (RHD-1) on HBV Carrier With Abnormal Liver Function: a Randomized Controlled Trial
Brief Title: The Effect of Compound Herbal Formula (RHD-1) on HBV Carrier With Abnormal Liver Function
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Taipei City Hospital (Other Government)
Collaborators: National Yang Ming Chiao Tung University (Other)
Responsible Party: Principal Investigator, Chung-Hua Hsu, vice president, Taipei City Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 100001-62-010; 100-00-62-01 (Other Grant/Funding Number: 100-00-62-01A)
Record Dates: First submitted 2011-04-18; First posted 2011-04-19 (Estimated); Last update posted 2014-05-07 (Estimated); Status verified 2014-05

CONDITIONS: Liver Dysfunction
Keywords: HBV carrier; HBV DNA title; Chinese Medicine; Liver function; RHD-1
MeSH Terms: conditions — Liver Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A foumula (Experimental): Compound Herbal Formula (RHD-1)
  Interventions: Other: Compound Herbal Formula (RHD-1)
- B formula (Placebo Comparator): dilute Compound Herbal Formula
  Interventions: Other: dilute RHD-1

INTERVENTIONS:
Other: Compound Herbal Formula (RHD-1) — 100 ml/per day
  Other Names: Chinese herbal medicine
  Arms: A foumula
Other: dilute RHD-1 — 100 ml/per day
  Other Names: Chinese herbal medicine dilute
  Arms: B formula

SUMMARY:
The aim of the study is to examine whether the compound herbal formula (RHD-1) is effective on HBV Carrier With Abnormal Liver Function.

DETAILED DESCRIPTION:
% change HBV DNA title and liver function.

ELIGIBILITY:
Inclusion Criteria:

* 40 < GPT <200 HBV carrier Age: 18-65 yrs old

Exclusion:

Creatinine >2.0 mg/dL Total bilirubin > 2.0mg/dL Not suitable patients diagnosis by physician in charge.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2011-05; Primary Completion 2012-06 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
the % change of HBV DNA title | 6 weeks

SECONDARY OUTCOMES:
the % change of GPT | 6 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei City Hospital, Taipei, Taiwan, Taiwan

REFERENCES:
- [Background] Hsu CH, Hwang KC, Chiang YH, Chou P. The mushroom Agaricus blazei Murill extract normalizes liver function in patients with chronic hepatitis B. J Altern Complement Med. 2008 Apr;14(3):299-301. doi: 10.1089/acm.2006.6344. PMID 18370584
- [Background] Chu CJ, Hussain M, Lok AS. Quantitative serum HBV DNA levels during different stages of chronic hepatitis B infection. Hepatology. 2002 Dec;36(6):1408-15. doi: 10.1053/jhep.2002.36949. PMID 12447866
- [Derived] Lee CJ, Cheng CH, Li YH, Liu CY, Hsu CH. A Chinese medicine, Kuan-Sin-Yin decoction, improves liver function in hepatitis B virus carriers: a randomized, controlled study. J Altern Complement Med. 2013 Dec;19(12):964-9. doi: 10.1089/acm.2013.0136. Epub 2013 Jul 17. PMID 23863086